CLINICAL TRIAL: NCT03511053
Title: Using Inflammatory Biomarkers and EMG Results to Predict Epidural Injection Response in Patients Diagnosed With Lumbar Stenosis
Brief Title: Epidural Lavage Study for Lumbar Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Thiru Annaswamy, Professor, PM&R, Principal Investigator, Staff Physician, Dallas VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-054
Record Dates: First submitted 2018-04-11; First posted 2018-04-27 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: Each participant receives a saline lavage followed by the lumbar epidural steroid injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Epidural Lavage followed by Lumbar Epidural Steroid Injection
  Interventions: Procedure: Epidural Steroid Injection with Lavage

INTERVENTIONS:
Procedure: Epidural Steroid Injection with Lavage — All participants will receive a saline lavage prior to the epidural steroid injection.

SUMMARY:
The purpose of this research is to find out if there are inflammatory biomarkers (also known as biological markers) in epidural space that can predict response to an epidural steroid injection. This study will also be evaluating whether the results of an EMG study (also known as electromyography) can predict the response to an epidural steroid injection.

DETAILED DESCRIPTION:
Lumbar spinal stenosis is a common cause of back pain and mobility impairment in older adults. It is often a multi-factorial condition resulting from degenerative changes in the spine, and may result in severe disability, with symptoms of lower back pain and/or pain, numbness and weakness of the lower extremities that are often exacerbated by walking and/or standing. Since lumbar spinal stenosis mostly stems from slowly progressive degenerative changes, symptoms often worsen over time, leading to poor health outcomes and high rates of healthcare utilization.

Epidural steroid injection (ESI) with anti-inflammatory compounds such as glucocorticoids is commonly provided to alleviate pain from neurogenic claudication in spinal stenosis: it is estimated that 25% of ESI's performed in the Medicare population and 74% of ESIs in the Veterans Affairs system are for spinal stenosis. However, one recent, large, multi-center, randomized controlled trial (RCT) demonstrated no significant benefit of epidural corticosteroids in alleviating symptoms of spinal stenosis. In this study, Friedly et al. conducted a double-blind, RCT comparing patient outcomes with epidural injection of glucocorticoid plus anesthetic (lidocaine) vs. anesthetic (lidocaine) only. No significant differences were observed at 6 weeks between the two groups of patients with respect to pain-related functional disability or pain intensity. However, a subset of patients who received glucocorticoids plus lidocaine reported significantly higher treatment satisfaction and higher reductions in depressive symptoms. This suggests that ESIs may be effective for a subset of patients with spinal stenosis.

Another treatment modality for spinal stenosis is decompression surgery, which may be effective for some patients but is associated with higher risk especially in the elderly and patients with multiple medical comorbidities. In Davis et al.'s observational study, in a two-year period with 68 patients, 32% of patients opted for surgery, 44% of patients were satisfied with non-surgical management and were discharged after 2 years, but the remaining 24% with non-surgical management (some of whom chose to decline surgery) did not seem to be satisfied with treatment. This study indicates the potential key role that non-surgical management options such as ESIs may play, in some patients. However, appropriate patient selection using indicators or biomarkers for patients who may most likely benefit from ESIs would be extremely beneficial.

In studying biomarkers that may predict patients' response to ESIs, Scuderi et al. found interferon-gamma (IFG) levels to have high predictive value for patients with lumbar nerve root irritation, while Golish et al. and Smith et al. found fibronectin-aggrecan complex (FAC) levels to have high predictive value for patients with herniated nucleus pulposus (HNP). In addition, many other factors (such as lower age and higher education) have been found to predict better outcome for radiculopathy. In particular, needle electromyography (EMG) has been shown in several studies to be a strong predictor for response to lumbar epidural steroid injection (LESI) and transforaminal epidural steroid injection (TESI) for patients with lumbosacral radiculopathy (LSR). Inspired by these studies, this study aims to explore if certain biomarkers such as IFG & FAC along with EMG findings can help predict which patients with spinal stenosis and neurogenic claudication will optimally benefit from ESIs.

ELIGIBILITY:
Inclusion Criteria:

* Mild-severe lumbar central canal stenosis identified by MRI or CT scan
* Symptoms:
* Lower extremety symptoms consistent with neurogenic claudication
* Pain, weakness and/or numbness triggered by standing or walking, and relieved by sitting
* Must be able to read English and complete assessment instruments

Exclusion Criteria:

* Cognitive impairment that renders the patient unable to give informed consent or provide accurate data
* Clinical co-morbidities that could interfere with the collection of data concerning pain and function
* Severe vascular, pulmonary, or coronary artery disease that limits ambulation including recent myocardial infarction (within 6 months)
* Spinal instability requiring surgical fusion
* Severe osteoporosis as defined by multiple compression fractures or a fracture at the same level as the stenosis
* Metastatic cancer
* Excessive alcohol consumption or evidence of non-prescribed or illegal drug use
* Pregnancy
* Concordant pain with internal rotation of the hip (or known hip joint pathology)
* Active local or systemic infection
* Abnormal coagulation
* Allergy to local anesthetic, steroid, or contrast
* Previous lumbar spine surgery
* Prisoners
* Epidural steroid injection within previous 6 months
* Rheumatological disorders such as rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thiru M Annaswamy, MD, Principal Investigator — Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrast MA. Epidural steroid injections for lumbar spinal stenosis. Curr Rev Musculoskelet Med. 2008 Mar;1(1):32-8. doi: 10.1007/s12178-007-9003-2. PMID 19468896
- [Background] Friedly JL, Bresnahan BW, Comstock B, Turner JA, Deyo RA, Sullivan SD, Heagerty P, Bauer Z, Nedeljkovic SS, Avins AL, Nerenz D, Jarvik JG. Study protocol- Lumbar Epidural steroid injections for Spinal Stenosis (LESS): a double-blind randomized controlled trial of epidural steroid injections for lumbar spinal stenosis among older adults. BMC Musculoskelet Disord. 2012 Mar 29;13:48. doi: 10.1186/1471-2474-13-48. PMID 22458343
- [Background] Friedly J, Nishio I, Bishop MJ, Maynard C. The relationship between repeated epidural steroid injections and subsequent opioid use and lumbar surgery. Arch Phys Med Rehabil. 2008 Jun;89(6):1011-5. doi: 10.1016/j.apmr.2007.10.037. PMID 18503793
- [Background] Friedly J, Chan L, Deyo R. Increases in lumbosacral injections in the Medicare population: 1994 to 2001. Spine (Phila Pa 1976). 2007 Jul 15;32(16):1754-60. doi: 10.1097/BRS.0b013e3180b9f96e. PMID 17632396
- [Background] Friedly JL, Comstock BA, Turner JA, Heagerty PJ, Deyo RA, Sullivan SD, Bauer Z, Bresnahan BW, Avins AL, Nedeljkovic SS, Nerenz DR, Standaert C, Kessler L, Akuthota V, Annaswamy T, Chen A, Diehn F, Firtch W, Gerges FJ, Gilligan C, Goldberg H, Kennedy DJ, Mandel S, Tyburski M, Sanders W, Sibell D, Smuck M, Wasan A, Won L, Jarvik JG. A randomized trial of epidural glucocorticoid injections for spinal stenosis. N Engl J Med. 2014 Jul 3;371(1):11-21. doi: 10.1056/NEJMoa1313265. PMID 24988555
- [Background] Suri P, Pashova H, Heagerty PJ, Jarvik JG, Turner JA, Bauer Z, Annaswamy TM, Nedeljkovic SS, Wasan AD, Friedly JL. Authors' Reply to Manchikanti. Spine (Phila Pa 1976). 2016 Feb;41(3):E183-4. doi: 10.1097/BRS.0000000000001142. No abstract available. PMID 26630434
- [Background] Davis N, Hourigan P, Clarke A. Transforaminal epidural steroid injection in lumbar spinal stenosis: an observational study with two-year follow-up. Br J Neurosurg. 2017 Apr;31(2):205-208. doi: 10.1080/02688697.2016.1206188. Epub 2016 Aug 22. PMID 27548310
- [Background] Scuderi GJ, Cuellar JM, Cuellar VG, Yeomans DC, Carragee EJ, Angst MS. Epidural interferon gamma-immunoreactivity: a biomarker for lumbar nerve root irritation. Spine (Phila Pa 1976). 2009 Oct 1;34(21):2311-7. doi: 10.1097/BRS.0b013e3181af06b6. PMID 19934811
- [Background] Golish SR, Hanna LS, Bowser RP, Montesano PX, Carragee EJ, Scuderi GJ. Outcome of lumbar epidural steroid injection is predicted by assay of a complex of fibronectin and aggrecan from epidural lavage. Spine (Phila Pa 1976). 2011 Aug 15;36(18):1464-9. doi: 10.1097/BRS.0b013e3181f40e88. PMID 21224775
- [Background] Smith MW, Ith A, Carragee EJ, Cheng I, Alamin TF, Golish SR, Mitsunaga K, Scuderi GJ, Smuck M. Does the presence of the fibronectin-aggrecan complex predict outcomes from lumbar discectomy for disc herniation? Spine J. 2019 Feb;19(2):e28-e33. doi: 10.1016/j.spinee.2013.06.064. Epub 2013 Nov 13. PMID 24239034
- [Background] Iversen T, Solberg TK, Wilsgaard T, Waterloo K, Brox JI, Ingebrigtsen T. Outcome prediction in chronic unilateral lumbar radiculopathy: prospective cohort study. BMC Musculoskelet Disord. 2015 Feb 7;16(1):17. doi: 10.1186/s12891-015-0474-9. PMID 25887469
- [Background] Annaswamy TM, Bierner SM, Chouteau W, Elliott AC. Needle electromyography predicts outcome after lumbar epidural steroid injection. Muscle Nerve. 2012 Mar;45(3):346-55. doi: 10.1002/mus.22320. PMID 22334168
- [Background] Fish DE, Shirazi EP, Pham Q. The use of electromyography to predict functional outcome following transforaminal epidural spinal injections for lumbar radiculopathy. J Pain. 2008 Jan;9(1):64-70. doi: 10.1016/j.jpain.2007.08.011. Epub 2007 Nov 5. PMID 17974488
- [Background] McCormick Z, Cushman D, Caldwell M, Marshall B, Ghannad L, Eng C, Patel J, Makovitch S, Chu SK, Babu AN, Walega DR, Marciniak C, Press J, Kennedy DJ, Plastaras C. Does Electrodiagnostic Confirmation of Radiculopathy Predict Pain Reduction after Transforaminal Epidural Steroid Injection? A Multicenter Study. J Nat Sci. 2015 Aug;1(8):e140. PMID 26251843
- [Result] Lin CK, Borresen A, Kroll M, Annaswamy TM. Predicting Response to Epidural Steroid Injections for Lumbar Spinal Stenosis with Biomarkers and Electromyography. PM R. 2020 Jul;12(7):663-670. doi: 10.1002/pmrj.12272. Epub 2019 Dec 28. PMID 31659847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Lumbar Spinal Stenosis were recruited from the spine clinic at the Veterans Affairs Medical Center, and were included in the study if they met the study criteria.
Period: Overall Study
Arm/Group | All Participants
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 11
Pain Disability Questionnaire [Mean (Full Range); unit: units on a scale] — The Pain Disability Questionnaire (PDQ) allows patients to rate their ability to complete specific tasks on a 10-cm visual analog scale (15 questions) ranging from having no problems with the task (zero) to being unable to complete it at all (ten).
  Psychosocial and functional component subscores and the total score are calculated based on the responses. The maximum total score is 150; the maximum psychosocial subscore is 60; and the maximum functional subscore is 90. Lower scores indicate less pain-related disability.
  units on a scale | 77.5 [64.6 to 90.4]
VAS-Questionnaires [Mean (Full Range); unit: units on a scale] — 0-10 visual analog scale. Lower numbers indicate lower levels of pain
  units on a scale | 64.1 [58.7 to 69.5]

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale
Description: Number rating of back/leg pain from 0 to 10, 0 being no pain/discomfort, 10 being extreme pain/discomfort
Time Frame: Change between baseline, 1 month and 2 months post injection
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 11
score on a scale
  Average at baseline | 6.2 [5.7 to 7]
  Average at 1 month | 5.0 [3.5 to 6.5]
  Average at 2 months | 5.0 [3.5 to 6.5]
  Average 1 month change | 0.8 [-0.8 to 2.4]
  Average 2 month change | 1 [-0.7 to 2.7]

2. Primary Outcome: Swiss Spinal Stenosis Questionnaire
Description: Measures how pain due to spinal stenosis is effected the patient based on quality of life/pain questions and satisfaction questions for months 1 and 2 (no scales are used) SSSQ scores are reported in percentages 0-100%, higher scores indicate worse outcomes.
Time Frame: Change between baseline, 1 month and 2 months post injection
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | All Participants
Number analyzed (Participants) | 11
Percentage
  Average at baseline | 64.1 [58.7 to 69.5]
  Average at 1 month | 53.2 [41.7 to 64.7]
  Average at 2 months | 53.5 [43.6 to 63.4]
  Average at 1 month change | 11.7 [-4.2 to 27.6]
  Average at 2 month change | 10.3 [-1.5 to 22.1]

3. Primary Outcome: Pain Disability Questionnaire
Description: Measures how pain is affecting the patients lifestyle on a scale from 0 to 10 as defined by each question. The questionnaire contains 15 questions that each range on a scale form 0 to 10. The total score of the questionnaire ranges from 0 to 150. Lower values represent a better outcome.
Time Frame: Change between baseline, 1 month and 2 months post injection
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 11
score on a scale
  Average at baseline | 77.5 [64.6 to 90.4]
  Average at 1 month | 53.3 [28.6 to 78]
  Average at 2 months | 64.3 [34.5 to 94.1]
  Average at 1 month change | 27.3 [7.6 to 47]
  Average at 2 month change | 16.2 [-10.2 to 42.6]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the day of consent for up to 16weeks, for each participant.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT03511053/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT03511053/ICF_001.pdf